CLINICAL TRIAL: NCT00506402
Title: A Phase 1 Study of MKC-1 in Patients With Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-104
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Hematological Malignancies; Myelodysplasia; Agnogenic Myeloid Metaplasia
Keywords: Adult patients with refractory leukemias, MDS or AMM
MeSH Terms: conditions — Hematologic Neoplasms; Anemia, Refractory, with Excess of Blasts; Primary Myelofibrosis

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MKC-1

INTERVENTIONS:
Drug: MKC-1 — Capsule, 30 mg and 100 mg, BID, continuous dosing

SUMMARY:
The main objectives of this study are to evaluate the side effects of MKC-1 and to determine a safe dose of MKC-1 for future studies in patients with hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have relapsed/refractory leukemias for which no standard therapies are anticipated to result in a durable remission. Patients with poor-risk myelodysplasia (MDS) [i.e. IPSS ≥ 1.5 or chronic myelomonocytic leukemia (CMML) are also candidates for this protocol. Relapsed/refractory leukemias include acute non-lymphocytic leukemia (AML) by WHO classification, acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blast crisis. Patients with agnogenic myeloid metaplasia (AMM) are also eligible.
2. Age > 18 years.
3. ECOG performance status of 0-2.
4. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents. If the patient is on hydroxyurea to control peripheral blood leukemic cell counts, the patient must be off hydroxyurea for at least 48 hours before initiation of treatment on this protocol.
5. Persistent clinically significant chronic toxicities from prior chemotherapy, surgery or radiotherapy must have resolved to NCI CTCAE Grade < 1, except for alopecia.
6. The following laboratory results, within 10 days of MKC-1 administration (unless the abnormality is considered attributable to leukemia):

   * Serum creatinine < 2.0 mg/dL
   * Total bilirubin < ULN (unless a diagnosis of Gilbert's disease is present)
   * AST < 2.5 x ULN (upper limit of normal)
   * Serum albumin > 3.0 g/dL
7. Signed informed consent.

Exclusion Criteria:

1. Pre-existing hepatomegaly with disease measured as > 2 cm below the costal margin, secondary to malignancy.
2. Pregnant or breast-feeding women. Female patients must be postmenopausal, surgically sterile or they must agree to use a physical method of contraception. Female patient with childbearing potential must have a negative pregnancy test within the 10 days before the first MKC-1 administration. Male patients must be surgically sterile or agree to use an acceptable method of contraception. Pregnant and nursing patients are excluded because the effects of MKC-1 on a fetus or nursing child are unknown.
3. Clinical evidence of bowel obstruction, active uncontrolled malabsorption syndromes or a history of total gastrectomy.
4. Impaired cardiac function including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure.
5. Patients receiving any other standard or investigational cytotoxic treatment for their hematologic malignancy.
6. Treatment with antiretroviral therapy metabolized through CYP3A4 (including indinavir, nelfinavir, ritonavir and saquinavir) due to the potential for drug interactions wth MKC-1.
7. Any medical conditions that, in the investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include congestive heart failure of Class III or IV of the NYHA classification, active infection, or any psychiatric condition that would interfere with the understanding of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events | Throughout study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yee, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Canada